CLINICAL TRIAL: NCT00937521
Title: A Phase 2 Partially Observer-Blind Randomized Controlled Multicenter Dose-Ranging and Formulation-Finding Study of a New Novartis Meningococcal B Recombinant Vaccine Evaluating the Safety and Immunogenicity When Given Concomitantly With Routine Vaccines in 2-month-old Infants
Brief Title: Safety and Immunogenicity in Dose-Ranging and Formulation-Finding Meningococcal B (MenB) Vaccine Study in 2-month-old Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V72P16; 2009-010106-11
Record Dates: First submitted 2009-06-29; First posted 2009-07-13 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Meningococcal Meningitis; Meningococcal Infections
Keywords: Immunogenicity; Meningitis; Antibody; Infants
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections; Meningitis | interventions — 4CMenB vaccine; Antipyretics

STUDY DESIGN:
Who Masked: Participant

ARMS (8):
- 1 (Other): Vaccine candidate formulation I
  Interventions: Biological: Meningococcal B vaccine
- 2 (Other): Vaccine candidate formulation II
  Interventions: Biological: Meningococcal B vaccine
- 3 (Other): Vaccine candidate formulation III
  Interventions: Biological: Meningococcal B vaccine
- 4 (Other): Vaccine candidate formulation IV
  Interventions: Biological: Meningococcal B vaccine
- 5 (Other): Vaccine candidate formulation V
  Interventions: Biological: Meningococcal B vaccine
- 6 (Other): Vaccine candidate formulation VI
  Interventions: Biological: Meningococcal B vaccine
- 7 (Other): Control
  Interventions: Biological: Control
- 8 (Other): Vaccine candidate formulation I with antipyretic
  Interventions: Biological: Meningococcal B vaccine with antipyretic

INTERVENTIONS:
Biological: Meningococcal B vaccine — Vaccine candidate formulation I
  Arms: 1
Biological: Meningococcal B vaccine — Vaccine candidate formulation II
  Arms: 2
Biological: Meningococcal B vaccine — Vaccine candidate formulation III
  Arms: 3
Biological: Meningococcal B vaccine — Vaccine candidate formulation IV
  Arms: 4
Biological: Meningococcal B vaccine — Vaccine candidate formulation V
  Arms: 5
Biological: Meningococcal B vaccine — Vaccine candidate formulation VI
  Arms: 6
Biological: Control — Control
  Arms: 7
Biological: Meningococcal B vaccine with antipyretic — Vaccine candidate formulation I with antipyretic
  Arms: 8

SUMMARY:
This study is aimed at assessing the safety and immunogenicity of different doses and formulations of a new Novartis Meningococcal B Recombinant Vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month old infants (55-89 days, inclusive), born after full term pregnancy, gestational age ≥ 37 weeks and a birth weight ≥ 2.5 kg
* Available for all the visits scheduled in the study and for whom a parent/legal guardian is willing/able to comply with all protocol requirements

Exclusion Criteria:

* Any meningococcal B or C vaccine administration
* Prior vaccination with any Diphtheria, Tetanus, Pertussis (acellular or whole cell), Polio (either Inactivated or Oral), Haemophilus influenzae type b (Hib), and Pneumococcal antigens;
* Any ascertained or suspected disease caused by N. meningitidis
* Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis
* History of severe allergic reaction after previous vaccinations
* Recent significant acute or chronic infection
* Oral or parenteral antibiotic treatment in the 7 days prior to the scheduled blood draw;
* Any serious chronic or progressive disease according to the judgment of the investigator (e.g., neoplasm, diabetes mellitus Type I, cardiac disease, hepatic disease, progressive neurological disease or seizure, either associated with fever or as part of an underlying neurological disorder or syndrome, autoimmune disease, HIV infection or AIDS, or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition)
* Any impairment/alteration of the immune system resulting from (for example):

  * Receipt of any immunosuppressive therapy at any time since birth
  * Receipt of immunostimulants at any time since birth
  * Use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids at any time since birth
* Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation
* Participation in another clinical trial
* Family members and household members of research staff
* History of seizure
* Any contraindication to paracetamol

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1507 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- Hospital Privado de Córdoba CMC SA, Naciones Unidas 346, Córdoba Province, Argentina
- Chile (2):
  - Universidad de Chile, Av Independencia 1027, Comuna de Independencia, Santiago Metropolitan
  - Consultorio Manuel Bustos, Lo Cruzat 486, Quilicura, Santiago Metropolitan
- Czechia (18):
  - Samostatna ordinace praktickeho lekare pro deti a dorost, O. Kubina 17, Boskovice
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Neklez 3, Brno
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Pernštýnská 127/l, Chlumec Nad Cidlinou
  - Zdravotní středisko, Vaclavska 4186, Chomutov
  - Nemocnice Decin, Detske oddělení, U Nemocnice 1, Děčín
  - Fakulta vojenskeho zdravotnictvi UO, Trebešská 1575, Hradec Králové
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Masarykova 389, Humpolec
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Ruských Legii 352, Jindřichův Hradec
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Hrnčířská 1401, Lipník Nad Bečvou
  - Oblastni nemocnice Nachod, Destske oddělení, Purkyňova 446, Náchod
  - Samostatna ordinace praktickeho lekare pro deti a dorost, U Lékárny 306, Odolena Voda
  - Prakticky lekar pro deti a dorost, Dvouletky 54, Ostrava
  - KHS Ostrava, Protiepidemické oddělení, Na Bělidle 7, Ostrava
  - Nemocnice Pardubice, Destske odděleni, Kyjevská 44, Pardubice
  - Fakultni nemocnice Bory, E. Beneše 13, Plzeň
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Chrudimska 2a, Praha 3
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Kladenská 53, Praha 6
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Velka Michalska 22, Znojmo
- Hungary (11):
  - Házi Gyermekorvosi szolgálat, Honvéd U.2., Bordány
  - Medszolg 2000 Bt, 6723, Szeged, Dandár u.4, Ányos U.4., Budapest
  - Erzsébet Kórház Gyermekosztály, Hódmezővásárhely, Dr. Imre József U.2.
  - Baby Box Bt,, 6724, Szeged, Kossuth Lajos sgt.109, Szeged, Kossuth Lajos Sgt.109
  - Dr. Bán Mariann és Társa Bt., Kando Kalman U.1, Miskolc
  - Futurnest Kft, Selyemrét U.1., Miskolc
  - Ped-Med Kft. , 3434 Mályi, Fő u.12., Fő U.12., Mályi
  - S.K. Sipka és Kovács Eü. Bt., Csongrádi Sgt. 63., Szeged
  - Oszila Kft. 6723, Szeged, Debreceni u.10-14., Debreceni U.10-14., Szeged
  - Győriné dr. Bari Eszter egyéni vállalkozó, Csongrád, Szentháromság Tér 10
  - Vas Megyei Markusovszky Kórház, Gyermekosztály, Markusovszky U. 1-3, Szombathely
- Italy (6):
  - Dipartimento di Neonatologia e Terapia Intensiva Neonatale, "Ospedale dei Bambini", Presidio Ospedaliero dell'Azienda Ospedaliera Spedali Civili di Brescia, P.le Spedali Di Brescia,1, Brescia
  - Dipartimento di Pediatria dell'Università degli Studi di Firenze, Viale Pieraccini N. 24, Firenze
  - Università degli Studi di Messina, Pad. NI - A.O.U. Policlinico G.Martino, Via Consolare Valeria, 1, Messina
  - Fondazione IRCCS dell'Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena di Milano, Via Commenda, 9, Milano
  - Pediatria dell'Ospedale Sacco di Milano, Via G.B.Grossi 74, Milano
  - Dipartimento di Pediatria Azienda Ospedaliera di Padova, Via Giustiniani, 3, Padova

REFERENCES:
- [Derived] Viviani V, Biolchi A, Pizza M. Synergistic activity of antibodies in the multicomponent 4CMenB vaccine. Expert Rev Vaccines. 2022 May;21(5):645-658. doi: 10.1080/14760584.2022.2050697. Epub 2022 Mar 14. PMID 35257644
- [Derived] Esposito S, Prymula R, Zuccotti GV, Xie F, Barone M, Dull PM, Toneatto D. A phase 2 randomized controlled trial of a multicomponent meningococcal serogroup B vaccine, 4CMenB, in infants (II). Hum Vaccin Immunother. 2014;10(7):2005-14. doi: 10.4161/hv.29218. PMID 25424810

RESULTS

PARTICIPANT FLOW:
Groups:
- B+OMV (Group I): Subjects in this group received one dose of meningococcal B recombinant (rMenB+OMV NZ) adsorbed vaccine (formulation I) and routine vaccines at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- B+½ OMV (Group II): Subjects in this group received one dose of meningococcal B recombinant (rMenB+OMV NZ) adsorbed vaccine (formulation II) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- B+1/4 OMV (Group III): Subjects in this group received one dose of meningococcal B recombinant (rMenB+OMV NZ) adsorbed vaccine (formulation III) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- B (Group IV): Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation IV) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- ½ (B+OMV) (Group V): Subjects in this group received one dose of meningococcal B recombinant (rMenB+OMV NZ) adsorbed vaccine (formulation V) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- PH2 B+OMV (Group VI): Subjects in this group received one dose of meningococcal B recombinant (rMenB+OMV NZ) adsorbed vaccine (formulation VI) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- MenC (Group VII): Subjects received one dose of meningococcal C conjugate vaccine (Menjugate®; Men C) and routine vaccine at 2,3,4 months of age, one dose of meningococcal B recombinant (rMenB+OMV NZ) adsorbed vaccine (formulation VII) and routine vaccine at 12 months of age, one dose of rMenB+OMV NZ and one dose of MenC at 13 months of age.
- Par+B+OMV (Group VIII): Subjects in this group received one dose of meningococcal B recombinant (rMenB+OMV NZ) adsorbed vaccine (formulation I) with paracetamol and routine vaccines at 2,3,4,12 months of age and MenCCRM197 at 13 months of age.
Period: Overall Study - Prior to Booster Dose
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Started | 188 | 190 | 192 | 188 | 191 | 188 | 186 | 184
Premature Withdrawal | 3 | 5 | 6 | 1 | 3 | 1 | 5 | 1
Completed | 185 | 185 | 186 | 187 | 188 | 187 | 181 | 183
Not Completed | 3 | 5 | 6 | 1 | 3 | 1 | 5 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 0 | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Inappropriate enrollment | 0 | 4 | 0 | 0 | 2 | 1 | 1 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Booster Phase
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Started | 155 | 163 | 169 | 170 | 168 | 165 | 165 | 161
Premature Withdrawal | 3 | 2 | 5 | 3 | 5 | 5 | 5 | 2
Completed | 152 | 161 | 164 | 167 | 163 | 160 | 160 | 159
Not Completed | 3 | 2 | 5 | 3 | 5 | 5 | 5 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 2 | 2 | 4 | 2 | 4 | 4 | 3 | 0
Not completed — Administrative Reason | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- B+OMV (Group I): Subjects in this group received one dose of meningococcal B recombinant adsorbed vaccine (formulation I) and routine vaccines at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- B+½ OMV (Group II): Subjects in this group received one dose of meningococcal B recombinant adsorbed vaccine (formulation II) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- B+1/4 OMV (Group III): Subjects in this group received one dose of meningococcal B recombinant adsorbed vaccine (formulation III) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- ½ (B+OMV) (Group V): Subjects in this group received one dose of meningococcal B recombinant adsorbed vaccine (formulation V) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- PH2 B+OMV (Group VI): Subjects in this group received one dose of meningococcal B recombinant adsorbed vaccine (formulation VI) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- Total: Total of all reporting groups
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII) | Total
Number analyzed (Participants) | 188 | 190 | 192 | 188 | 191 | 188 | 186 | 184 | 1507
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 188 | 190 | 192 | 188 | 191 | 188 | 186 | 184 | 1507
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 91 | 82 | 96 | 79 | 93 | 98 | 72 | 699
  Male | 100 | 99 | 110 | 92 | 112 | 95 | 88 | 112 | 808

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Serum Bactericidal Activity (hSBA) ≥ 1:5 at 1 Month After Third Vaccination
Description: To assess the immunogenicity of seven different formulations of 4CMenB (groups I-VI and VIII) given to healthy infants at 2,3 and 4 months of age as measured by percentages of subjects with serum bactericidal activity (SBA) titer≥1:5 against 44/76-SL, 5/99 and NZ98/254 reference strains, at 1 month after the third vaccination.. The analysis was done on the Per Protocol Primary Population at one month after third injection.
Time Frame: At baseline (pre-vaccination) and 30 days after the third vaccination.
Population: Analysis as per PP population.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 171 | 174 | 171 | 174 | 172 | 173 | 171 | 169
Percentages of Subjects
  44/76SLBaseline(N=166,171,168,170,169,168,168,166) | 5 [2 to 9] | 2 [0 to 5] | 4 [1 to 8] | 4 [2 to 8] | 4 [2 to 8] | 4 [2 to 8] | 2 [1 to 6] | 3 [1 to 7]
  44/76-SL > 3rd(N=170,170,166,166,169,167,165,167) | 100 [98 to 100] | 99 [97 to 100] | 99 [97 to 100] | 100 [98 to 100] | 99 [97 to 100] | 99 [96 to 100] | 6 [3 to 11] | 100 [98 to 100]
  5/99-Baseline (N=162,162,161,161,166,166,161,157) | 5 [2 to 9] | 3 [1 to 7] | 6 [3 to 10] | 4 [2 to 9] | 8 [5 to 14] | 4 [2 to 8] | 6 [3 to 10] | 4 [1 to 8]
  5/99 > 3rd (N=165,167,161,166,165,161,159,160) | 99 [97 to 100] | 100 [98 to 100] | 99 [97 to 100] | 100 [98 to 100] | 100 [98 to 100] | 99 [97 to 100] | 3 [1 to 7] | 99 [97 to 100]
  NZ98/254Baseline(N=170,174,171,174,171,173,171,169 | 1 [0.015 to 3] | 0 [0 to 2] | 1 [0.015 to 3] | 1 [0.015 to 3] | 1 [0 to 4] | 1 [0 to 4] | 2 [0 to 5] | 1 [0.015 to 3]
  NZ98/254 > 3rd (N=171,172,169,168,172,169,168,168) | 78 [71 to 84] | 67 [59 to 74] | 56 [48 to 64] | 1 [0.015 to 3] | 62 [54 to 69] | 81 [74 to 87] | 2 [0 to 5] | 74 [67 to 81]

2. Secondary Outcome: Geometric Mean Bactericidal Titers (GMTs), One Month After Third and Booster Vaccination (Men B at 12 Months of Age)
Description: ToTo assess the immune response of seven different formulations of meningococcal multi-component recombinant, adsorbed vaccine (rMenB+OMV NZ or rMenB (no OMV)) in healthy toddlers as measured by SBA geometric mean titers (GMTs) at:
  1. One month after third vaccination.
  2. One month after booster vaccination (Men B at 12 months of age).
Time Frame: At baseline (pre-vaccination), 30 days after the third vaccination, at booster Baseline and at booster vaccination (12 months of age)
Population: Per Protocol Primary and Booster populations.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 171 | 174 | 171 | 174 | 172 | 173 | 171 | 169
Titers
  44/76-SL Base(N=166,171,168,170,169,168,168,166) | 1.25 [1.14 to 1.37] | 1.12 [1.03 to 1.23] | 1.2 [1.1 to 1.32] | 1.19 [1.08 to 1.3] | 1.31 [1.19 to 1.43] | 1.2 [1.09 to 1.31] | 1.16 [1.09 to 1.25] | 1.18 [1.08 to 1.3]
  44/76-SL > 3(N=170,170,166,166,169,167,165,167) | 101 [90 to 113] | 112 [101 to 126] | 113 [101 to 126] | 62 [56 to 70] | 71 [64 to 80] | 102 [92 to 114] | 1.24 [1.11 to 1.39] | 102 [91 to 115]
  44/76-SL - Base Boost(N=69,78,74,78,71,71,74,70) | 4.94 [3.76 to 6.5] | 5.22 [4.03 to 6.76] | 5.72 [4.41 to 7.42] | 5.44 [4.19 to 7.06] | 3.96 [3.02 to 5.18] | 3.76 [2.87 to 4.94] | 1.15 [1.03 to 1.29] | 4.51 [3.43 to 5.95]
  44/76-SL > Boost(N=65,73,70,75,76,71,75,63) | 120 [95 to 150] | 152 [122 to 189] | 118 [95 to 146] | 53 [43 to 66] | 99 [79 to 122] | 105 [84 to 131] | 12 [10 to 16] | 136 [107 to 172]
  5/99-Baseline-(N=162,162,161,161,166,166,161,157) | 1.18 [1.07 to 1.3] | 1.09 [0.99 to 1.2] | 1.12 [1.02 to 1.23] | 1.13 [1.03 to 1.25] | 1.3 [1.18 to 1.43] | 1.16 [1.05 to 1.27] | 1.21 [1.09 to 1.34] | 1.07 [0.97 to 1.18]
  5/99 > 3 (N=165,167,161,166,165,161,160) | 396 [348 to 450] | 503 [442 to 572] | 534 [469 to 608] | 389 [342 to 443] | 316 [278 to 360] | 371 [326 to 422] | 1.15 [1.03 to 1.29] | 455 [399 to 519]
  5/99 Base Boost(N=71,76,80,72,77,78,70,71) | 69 [53 to 88] | 91 [71 to 116] | 111 [87 to 141] | 74 [57 to 94] | 54 [42 to 68] | 64 [50 to 81] | 1.11 [0.95 to 1.29] | 106 [82 to 136]
  5/99 > Boost(N=73,77,79,72,76,74,69,76) | 1950 [1573 to 2417] | 1819 [1478 to 2238] | 2238 [1820 to 2751] | 730 [590 to 903] | 983 [801 to 1205] | 1321 [1074 to 1624] | 41 [29 to 57] | 2182 [1769 to 2691]
  NZ98/254-BaselineN=170,174,171,174,171,173,171,169 | 1.02 [0.99 to 1.06] | 1.02 [0.99 to 1.05] | 1.03 [1 to 1.06] | 1.04 [1 to 1.07] | 1.03 [1 to 1.06] | 1.04 [1.01 to 1.08] | 1.06 [1 to 1.13] | 1.02 [0.99 to 1.05]
  1month after 3rd vaccN=171,172,169,172,169,169,168 | 10 [8.59 to 12] | 7.81 [6.69 to 9.12] | 5.74 [4.92 to 6.71] | 1.05 [0.9 to 1.23] | 6.66 [5.71 to 7.77] | 11 [9.16 to 13] | 1.05 [1.01 to 1.1] | 8.48 [7.24 to 9.93]
  NZ98/254 Bas Bst N=141,155,155,150,150,153,148,143 | 1.6 [1.43 to 1.8] | 1.28 [1.15 to 1.43] | 1.23 [1.1 to 1.37] | 1.11 [0.99 to 1.24] | 1.35 [1.21 to 1.5] | 1.41 [1.26 to 1.57] | 1.03 [1 to 1.06] | 1.48 [1.32 to 1.66]
  1month after boosterN=138,152,150,149,152,146,140 | 20 [16 to 24] | 18 [15 to 22] | 11 [9.07 to 13] | 1.67 [1.38 to 2.03] | 14 [12 to 17] | 20 [16 to 24] | 2.2 [1.89 to 2.57] | 20 [17 to 25]

3. Secondary Outcome: Geometric Mean Bactericidal Titers,One Month After Primary and Booster Vaccination (Men B at 12 Months of Age)
Description: To compare the antibody response of meningococcal multi-component recombinant, adsorbed vaccine (formulation I vs. formulation VIII) and of routine infant vaccine given with or without prophylactic administration of paracetamol medication in healthy toddlers.
Time Frame: At Baseline (pre-vaccination), at 30 days after the third vaccination, at booster Baseline, at 30 days
Population: As per PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+OMV (Group I) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 171 | 169
Titers
  44/76-SL Strain - Baseline (N=166,166) | 1.25 [1.14 to 1.37] | 1.18 [1.08 to 1.3]
  44/76-SL > 3rd (N=170,167) | 101 [90 to 113] | 102 [91 to 115]
  44/76-SL Baseline booster (N=69,70) | 4.94 [3.76 to 6.5] | 4.51 [3.43 to 5.95]
  44/76-SL > booster (N=65,63) | 120 [95 to 150] | 136 [107 to 172]
  5/99 Strain - Baseline (N=162,157) | 1.18 [1.07 to 1.3] | 1.07 [0.97 to 1.18]
  5/99 > 3rd (N=165,160) | 396 [348 to 450] | 455 [399 to 519]
  5/99 Baseline booster (N=71,71) | 69 [53 to 88] | 106 [82 to 136]
  5/99 > booser (N=73,76) | 1950 [1573 to 2417] | 2182 [1769 to 2691]
  NZ98/254 Strain-Baseline (N=170,169) | 1.02 [0.99 to 1.06] | 1.02 [0.99 to 1.05]
  NZ98/254 > 3rd (N=171,168) | 10 [8.59 to 12] | 8.48 [7.24 to 9.93]
  NZ98/254 Baseline booster (N=141,143) | 1.6 [1.43 to 1.8] | 1.48 [1.32 to 1.66]
  NZ98/254 > booster (N= 138, 140) | 20 [16 to 24] | 20 [17 to 25]

4. Secondary Outcome: Geometric Mean Ratios, One Month After Primary and Booster Vaccination (Men B at 12 Months of Age)
Description: To compare the antibody response between meningococcal multi-component recombinant adsorbed vaccine (formulation I) and routine infant vaccine group along with meningococcal multi-component recombinant adsorbed vaccine with prophylactic administration of paracetamol medication as measured by Geometric Mean Ratios (GMRs).
Time Frame: After the third and the booster vaccination.
Population: As per PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | B+OMV (Group I) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 162 | 160
Ratios
  44/76-SL > 3rd (N=157,157) | 80 [69 to 93] | 84 [72 to 97]
  44/76-SL > Booster (N=59,56) | 24 [18 to 31] | 28 [21 to 36]
  5/99 > 3rd (N=152,142) | 345 [292 to 408] | 417 [350 to 497]
  5/99 > Booster (N=68,68) | 27 [21 to 35] | 20 [16 to 25]
  NZ98/254 > 3rd (N=162,160) | 9.65 [8.19 to 11] | 8.69 [7.36 to 10]
  NZ98/254 > Booster (N=129,127) | 12 [10 to 15] | 14 [11 to 17]

5. Secondary Outcome: Percentage of Subjects With hSBA≥1:5, Persistence of Bactericidal Antibodies at 12 Months of Age (Pre-fourth Dose)
Description: To assess the persistence of bactericidal antibodies at 12 months of age after primary vaccination - three doses of one of the seven different formulations of rMenB+OMV NZ or rMenB (no OMV) (Group I-VI and VIII) and rMenB+OMV NZ with paracetamol medication.
Time Frame: 12 months (pre-fourth vaccination)
Population: The analysis was done on the Per Protocol Booster population.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 141 | 155 | 155 | 150 | 150 | 153 | 148 | 143
Percentages of Subjects
  44/76-SL Pre-Boost(N=69,78,74,78,71,71,74,70) | 55 [43 to 67] | 58 [46 to 69] | 66 [54 to 77] | 63 [51 to 74] | 45 [33 to 57] | 44 [32 to 56] | 4 [1 to 11] | 47 [35 to 59]
  5/99 Pre-Boost(N=71,76,80,72,77,78,70,71) | 97 [90 to 100] | 100 [95 to 100] | 100 [95 to 100] | 97 [90 to 100] | 97 [91 to 100] | 99 [93 to 100] | 1 [0.036 to 8] | 100 [95 to 100]
  NZ98/254 Pre-B(N=141,155,155,150,150,153,148,143) | 12 [7 to 19] | 6 [3 to 11] | 5 [2 to 10] | 3 [1 to 7] | 7 [3 to 12] | 8 [4 to 13] | 0 [0 to 2] | 11 [7 to 18]

6. Secondary Outcome: Percentage of Subjects With hSBA≥1:5, Persistence of Bactericidal Antibodies at 12 Months of Age (One Month-post Fourth Dose)
Description: To assess if any of seven different formulations of rMenB+OMV NZ or rMenB (no OMV) vaccine (groups I-VI and VIII) induced sufficient immune response when given to healthy toddlers at 12 months of age, as measured by percentage of subjects with SBA titer ≥ 1:5, at 1 month after the fourth vaccination.
Time Frame: 1 month after fourth vaccination
Population: The analysis was done on the Per Protocol Booster population.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 138 | 152 | 150 | 149 | 152 | 146 | 147 | 140
Percentages of Subjects
  44/76-SL > Booster(N=65,73,70,75,76,71,63) | 100 [94 to 100] | 100 [95 to 100] | 100 [95 to 100] | 97 [91 to 100] | 100 [95 to 100] | 99 [92 to 100] | 84 [74 to 91] | 100 [94 to 100]
  5/99 strain (N=73,77,79,72,76,74,76) | 100 [95 to 100] | 100 [95 to 100] | 100 [95 to 100] | 100 [95 to 100] | 100 [95 to 100] | 100 [95 to 100] | 93 [84 to 98] | 100 [95 to 100]
  NZ98/254 (N=138,152,150,149,152,146,147,140) | 89 [83 to 94] | 89 [83 to 93] | 78 [71 to 84] | 18 [12 to 25] | 83 [76 to 89] | 88 [82 to 93] | 24 [18 to 32] | 90 [84 to 94]

7. Secondary Outcome: Geometric Mean Bactericidal Titers, After Primary and Booster Vaccinations (Men B at 12 Months of Age)
Description: To assess the induction of immunological memory of three doses of meningococcal multi-component recombinant, adsorbed vaccine by comparing the serum bactericidal antibodies Geometric Mean Bactericidal Titers (GMTs) response in healthy toddlers administered the fourth dose at 12 months of age to the response in meningococcal B vaccine naive toddlers (Group VII) receiving the first dose of meningococcal multi-component recombinant, adsorbed vaccine at 12 months of age.
Time Frame: At 13 months
Population: The analysis was done on the Per Protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+OMV (Group I) | MenC (Group VII)
Number analyzed (Participants) | 138 | 147
Titers
  44/76-SL > Booster (N=65,75) | 120 [95 to 150] | 12 [10 to 16]
  5/99 > Booster (N=73,69) | 1950 [1573 to 2417] | 41 [29 to 57]
  NZ98/254 > Booster | 20 [16 to 24] | 2.2 [1.89 to 2.57]

8. Secondary Outcome: Percentage of Subjects With hSBA ≥1:5, First Dose of Meningococcal B Vaccine (One Month After Booster)
Description: To assess the immune response of first dose of meningococcal multi-component recombinant, adsorbed vaccine given at 12 months of age to toddlers who previously received three doses of MenC-CRM197 vaccine as infants (group VII).
Time Frame: 1 month after booster
Population: The analysis was done on the Per Protocol population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | MenC (Group VII)
Number analyzed (Participants) | 147
Percentage of Subjects
  44/76-SL > Booster (N=75) | 84 [74 to 91]
  5/99 > Booster (N=69) | 93 [84 to 98]
  NZ98/254 > Booster | 24 [18 to 32]

9. Secondary Outcome: Safety and Reactogenicity of Study Vaccines Within 7 Days After Second and Third Vaccination
Description: To assess if any of six different formulations of rMenB+OMV NZ or rMenB (no OMV) vaccine (Group II to VI, Group VIII) reduced the incidence of fever ≥ 38.5ºC (rectal) occurring within 3 days (day 1-3) following second and third vaccination and 7 days (day 1-7) following each vaccination as compared to rMenB+OMV NZ (Group I).
Time Frame: Day 1 through day 7 after second and third vaccination.
Population: As per safety dataset.
Measure: Number; unit: Subjects
Groups:
- ½ (B+OMV) (Group V): Subjects in this group received one dose of meningococcal multi-component recombinant, adsorbed vaccine (formulation V)and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 182 | 180 | 186 | 184 | 182 | 180 | 177 | 179
Subjects
  Second Vaccination (day1-3) | 90 | 82 | 76 | 35 | 74 | 89 | 30 | 33
  3rd vac d 1-3(N=181,179,185,183,181,180,177,179) | 55 | 50 | 36 | 15 | 40 | 53 | 12 | 20
  First Vaccination (day1-7) | 94 | 91 | 74 | 24 | 60 | 76 | 22 | 46
  Second Vaccination (day 1-7) | 90 | 82 | 77 | 36 | 74 | 90 | 30 | 35
  3rd vac d 1-7(N=181,179,185,183,181,180,177,179) | 55 | 53 | 38 | 16 | 42 | 54 | 14 | 20
  Booster d 1-7(N=155,162,169,168,168,165,164,159) | 81 | 86 | 64 | 43 | 78 | 68 | 84 | 58

10. Secondary Outcome: Number of Subjects With Solicited Local Reactions Within 7 Days (Day 1-7) After Each Vaccination
Description: To assess the safety and tolerability of each of seven different formulations of rMenB+OMV NZ or rMenB (no OMV) vaccine (group I to VI, group VIII) in terms of number of subjects reporting solicited local reactions within 7 days (day 1-7) after each vaccination.
Time Frame: Day 1 through day 7 after each vaccination.
Population: The analysis was performed on the safety population.
Measure: Number; unit: Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 182 | 180 | 186 | 184 | 182 | 180 | 177 | 179
Subjects
  Any Local (First Vacc) | 163 | 155 | 153 | 123 | 141 | 157 | 127 | 137
  Injection Site Tenderness (First Vacc) | 114 | 116 | 111 | 54 | 97 | 121 | 48 | 79
  Injection Site Erythema (First Vacc) | 108 | 99 | 94 | 53 | 77 | 106 | 45 | 73
  Injection Site Induration (First Vacc) | 101 | 98 | 85 | 48 | 86 | 84 | 25 | 82
  Injection Site Swelling (First Vacc) | 58 | 49 | 55 | 24 | 48 | 60 | 15 | 41
  Any Local (Second Vacc) | 156 | 156 | 155 | 126 | 132 | 156 | 118 | 140
  Injection Site Tenderness (Second Vacc) | 121 | 116 | 97 | 48 | 88 | 116 | 47 | 85
  Injection Site Erythema (Second Vacc) | 104 | 114 | 114 | 71 | 90 | 104 | 44 | 94
  Injection Site Induration (Second Vacc) | 103 | 105 | 97 | 63 | 83 | 94 | 38 | 79
  Injection Site Swelling (Second Vacc) | 64 | 61 | 54 | 34 | 50 | 58 | 21 | 52
  Any Local (3rd N=181,179,185,183,181,180,177,179) | 151 | 147 | 141 | 122 | 130 | 152 | 113 | 128
  Injection Site Tenderness (Third Vacc) | 102 | 98 | 78 | 47 | 77 | 111 | 42 | 66
  Injection Site Erythema (Third Vacc) | 110 | 106 | 112 | 72 | 94 | 101 | 63 | 91
  Injection Site Induration (Third Vacc) | 97 | 92 | 92 | 62 | 79 | 89 | 55 | 80
  Injection Site Swelling (Third Vacc) | 56 | 56 | 46 | 35 | 45 | 58 | 29 | 47
  Any Local BoostN=155,162,169,168,168,165,162,159 | 131 | 132 | 149 | 113 | 127 | 130 | 133 | 121
  Injection Site Tenderness (Booster Vacc) | 116 | 107 | 120 | 77 | 106 | 112 | 108 | 92
  Injection Site Erythema (Booster Vacc) | 90 | 101 | 116 | 67 | 80 | 85 | 93 | 81
  Injection Site Induration (Booster Vacc) | 73 | 83 | 95 | 56 | 66 | 73 | 62 | 60
  Injection Site Swelling (Booster Vacc) | 55 | 59 | 69 | 31 | 47 | 52 | 39 | 47

11. Primary Outcome: Number of Subjects With Fever ≥ 38.5 °C (Rectal Temperature) Within 3 Days (Day 1-3) After First Vaccination
Description: To assess if any of six different formulations of vaccine groups (Group II to Group VI, Group VIII) reduced the incidence of fever >=38.5C (rectal) occurring within three days (day 1-day3) following first vaccination. The analysis was done on the Safety Population.
Time Frame: Day 1 to day 3 after first vaccination.
Population: The analysis was done on the Safety Population.
Measure: Number; unit: Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 182 | 180 | 186 | 184 | 182 | 180 | 177 | 179
Subjects | 94 | 91 | 74 | 24 | 60 | 76 | 21 | 46

12. Secondary Outcome: Number of Subjects With Solicited Systemic Reactions Within 7 Days (Day 1-7) After Each Vaccination
Description: To assess the safety and tolerability of each of seven different formulations of rMenB+OMV NZ or rMenB (no OMV) vaccine (group I to VI, group VIII) in terms of number of subjects reporting solicited systemic reactions within 7 days (day 1-7) after each vaccination.
Time Frame: Day 1 through day 7 after each vaccination.
Population: The analysis was performed on the safety population.
Measure: Number; unit: Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 182 | 180 | 186 | 184 | 182 | 180 | 177 | 179
Subjects
  Any Systemic (First Vacc) | 167 | 173 | 175 | 152 | 162 | 171 | 136 | 150
  Change Eat. Habits (First Vacc) | 76 | 87 | 84 | 52 | 84 | 90 | 41 | 66
  Sleepiness (First Vacc) | 120 | 131 | 119 | 96 | 117 | 119 | 92 | 116
  Vomiting (First Vacc) | 24 | 18 | 25 | 15 | 22 | 26 | 17 | 22
  Diarrhea (First Vacc) | 57 | 55 | 54 | 31 | 41 | 49 | 45 | 41
  Irritability (First Vacc) | 128 | 124 | 128 | 99 | 131 | 131 | 79 | 97
  Unus Crying (First Vacc) | 95 | 101 | 105 | 61 | 96 | 108 | 63 | 74
  Rash (First Vacc) | 6 | 5 | 5 | 7 | 10 | 10 | 4 | 5
  Fever ( ≥ 38.5°C ) (First Vacc) | 94 | 91 | 74 | 24 | 60 | 76 | 22 | 46
  Antipyr. Med. Used (First Vacc) | 102 | 94 | 92 | 37 | 74 | 95 | 32 | 166
  Any Systemic (Second Vacc) | 168 | 158 | 166 | 144 | 156 | 158 | 126 | 147
  Change Eat. Habits (Second Vacc) | 62 | 55 | 58 | 53 | 60 | 80 | 33 | 54
  Sleepiness (Second Vacc) | 105 | 100 | 102 | 85 | 92 | 109 | 75 | 84
  Vomiting (Second Vacc) | 18 | 18 | 14 | 15 | 17 | 20 | 14 | 20
  Diarrhea (Second Vacc) | 43 | 41 | 47 | 40 | 39 | 47 | 39 | 40
  Irritability (Second Vacc) | 130 | 121 | 124 | 94 | 117 | 126 | 82 | 99
  Unus Crying (Second Vacc) | 90 | 90 | 84 | 70 | 83 | 99 | 45 | 71
  Rash (Second Vacc) | 4 | 9 | 4 | 5 | 7 | 4 | 5 | 5
  Fever ( ≥ 38.5°C ) (Second Vacc) | 90 | 82 | 77 | 36 | 74 | 90 | 30 | 35
  Antipyr. Med. Used (Second Vacc) | 100 | 94 | 83 | 40 | 79 | 105 | 39 | 163
  Any Syst (3rdN=181,179,185,182,181,180,177,179) | 146 | 131 | 132 | 122 | 141 | 151 | 106 | 127
  Change Eat. Habits (Third Vacc) | 49 | 50 | 42 | 37 | 45 | 60 | 22 | 48
  Sleepiness (Third Vacc) | 75 | 67 | 82 | 64 | 77 | 79 | 52 | 75
  Vomiting (Third Vacc) | 8 | 18 | 15 | 12 | 12 | 13 | 11 | 20
  Diarrhea (Third Vacc) | 33 | 29 | 39 | 31 | 34 | 40 | 19 | 32
  Irritability (Third Vacc) | 115 | 97 | 93 | 74 | 104 | 115 | 76 | 84
  Unus Crying (Third Vacc) | 76 | 82 | 62 | 47 | 69 | 100 | 38 | 47
  Rash (Third Vacc) | 1 | 6 | 4 | 2 | 8 | 10 | 6 | 6
  Fever ( ≥ 38.5°C ) (Third Vacc) | 55 | 53 | 38 | 16 | 42 | 54 | 14 | 20
  Antipyr. Med. Used (Third Vacc) | 66 | 60 | 51 | 26 | 49 | 63 | 20 | 153
  Any Syst(BoosterN=155,162,169,169,168,165,164,159) | 143 | 144 | 139 | 118 | 141 | 142 | 142 | 137
  Change Eat. Habits (Booster Vacc) | 74 | 77 | 79 | 52 | 70 | 80 | 59 | 66
  Sleepiness (Booster Vacc) | 76 | 90 | 90 | 63 | 86 | 88 | 85 | 80
  Vomiting (Booster Vacc) | 6 | 11 | 7 | 7 | 10 | 9 | 9 | 20
  Diarrhea (Booster Vacc) | 30 | 34 | 36 | 43 | 32 | 30 | 26 | 30
  Irritability (Booster Vacc) | 116 | 111 | 112 | 86 | 116 | 115 | 117 | 96
  Unus Crying (Booster Vacc) | 74 | 64 | 69 | 46 | 71 | 82 | 73 | 50
  Rash (Booster Vacc) | 5 | 5 | 8 | 2 | 8 | 4 | 6 | 5
  Fever ( ≥ 38.5°C ) (Booster Vacc) | 81 | 86 | 64 | 43 | 78 | 68 | 84 | 58
  Antipyr. Med. Used (Booster Vacc) | 84 | 82 | 83 | 42 | 75 | 80 | 92 | 128

13. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events Within 7 Days (Day 1-7) After Each Vaccination
Description: To assess the safety and tolerability of each of seven different formulations of rMenB+OMV NZ or rMenB (no OMV) vaccine (group I to VI, group VIII) in terms of number of subjects reporting unsolicited Adverse Events (AEs), serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal (throughout the study period) within 7 days (day 1-7) after each vaccination.
Time Frame: Day 1 through day 7 after each vaccination.
Population: The analysis was performed on the safety population.
Measure: Number; unit: Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 184 | 184 | 189 | 187 | 187 | 185 | 184 | 183
Subjects
  Any AE (Day 1 to 7) (First Vacc) | 55 | 52 | 51 | 33 | 35 | 39 | 27 | 42
  At least Possibly related AE (First Vacc) | 48 | 48 | 43 | 30 | 27 | 34 | 22 | 36
  Any SAE (First Vacc) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Any AE D1-7 2nd N=182,181,186,184,183,180,178,180 | 55 | 53 | 50 | 41 | 36 | 47 | 28 | 45
  At least Possibly related AE (Second Vaccination) | 49 | 45 | 45 | 36 | 33 | 41 | 26 | 39
  Any SAE (Second Vacc) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Any AE D1-7 3rd N=182,181,186,184,182,180,177,179 | 40 | 59 | 49 | 35 | 31 | 45 | 35 | 39
  At least Possibly related AE (Third Vacc) | 34 | 52 | 45 | 29 | 23 | 37 | 29 | 36
  Any SAE (Third Vacc) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Any AE D 1-7Boos N=155,163,169,169,168,165,165,161 | 35 | 46 | 56 | 35 | 29 | 30 | 37 | 30
  At least Possibly related AE (Booster Vacc) | 28 | 41 | 48 | 23 | 23 | 26 | 30 | 25
  Any SAE (Booster Vacc) | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0

14. Secondary Outcome: Number of Subjects With Severe Adverse Events and Adverse Events Necessitating a Medical Office or Emergency Room (ER) Visit and/or Resulting in Premature Withdrawal of the Subject From the Study, Throughout the Study Period.
Description: To assess the safety and tolerability of each of seven different formulations of rMenB+OMV NZ or rMenB (no OMV) vaccine (group I to VI, group VIII) in terms of number of subjects reporting Severe Adverse Events (SAEs) and Adverse Events (AEs) necessitating a medical office or Emergency Room (ER) visit and/or resulting in premature withdrawal of the subject from the study, throughout the study period.
Time Frame: Overall study period.
Population: The analysis was performed on the safety population.
Measure: Number; unit: Subjects
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII)
Number analyzed (Participants) | 184 | 184 | 189 | 187 | 187 | 185 | 184 | 183
Subjects
  AE Leading to Premature Withdrawal-Primary Vacc | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 1
  Treatment Emergent SAEs - Primary Vacc | 16 | 20 | 12 | 20 | 13 | 16 | 11 | 15
  Tr E SAE Boost (N=155,163,169,169,168,165,165,161) | 14 | 7 | 12 | 5 | 15 | 9 | 9 | 16

15. Secondary Outcome: Number of Subjects With Local and Systemic Reactions Within 7 Days (Day 1-7) After Second rMenB+OMV NZ Vaccination in MenC Group
Description: To assess the safety and tolerability of two doses of rMenB+OMV NZ vaccine (Group VII) given at 12 and 13 months of age to toddlers who previously received three doses of Menjugate as infants.
Time Frame: Day 1 through day 7 at 13 months age.
Population: The analysis was performed on the safety population.
Measure: Number; unit: Subjects
Arm/Group | MenC (Group VII)
Number analyzed (Participants) | 156
Subjects
  Injection Site Tenderness | 92
  Injection Site Erythema | 84
  Injection Site Induration | 59
  Injection Site Swelling | 35
  Change Eat. Habits (N=155) | 43
  Sleepiness | 57
  Vomiting | 8
  Diarrhea | 18
  Irritability | 75
  Unus Crying | 37
  Rash | 4
  Fever ( ≥ 38.5°C ) (N=158) | 35
  Antipyr. Med. Used (N=157) | 47

ADVERSE EVENTS:
Time Frame: All solicited AEs and unsolicited AEs were collected from Day 1 to Day 7; serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal were collected during the overall study period.
Groups:
- B+OMV (Group I): Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation I) and routine vaccines at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to be applicable Prior to Booster Phase for AEs reporting.
- B+½ OMV (Group II): Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation II) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to be applicable Prior to Booster Phase for AEs reporting.
- B+1/4 OMV (Group III): Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation III) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to be applicable Prior to Booster Phase for AEs reporting.
- B (Group IV): Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation IV) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to be applicable Prior to Booster Phase for AEs reporting..
- ½ (B+OMV) (Group V): Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation V) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to be applicable Prior to Booster Phase for AEs reporting.
- PH2 B+OMV (Group VI): SubjSubjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation VI) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to be applicable Prior to Booster Phase for AEs reporting.
- MenC (Group VII): Subjects received one dose of meningococcal C conjugate vaccine (Menjugate®; Men C) and routine vaccine at 2,3,4 months of age and one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation VII) and routine vaccine at 12 months of age. One dose of MenC at 13 months of age.
  Group defined to be applicable Prior to Booster Phase for AEs reporting.
- Par+B+OMV (Group VIII): Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation I) with paracetamol and routine vaccines at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age. Group defined to be applicable Prior to Booster Phase for AEs reporting.
- B+OMV (Group I) Booster Phase: Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation I) and routine vaccines at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
- B+½ OMV (Group II) Booster Phase: Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine(formulation II) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to include Booster Phase.
- B+1/4 OMV (Group III) Booster Phase: Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation III) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to include Booster Phase.
- B (Group IV) Booster Phase: Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation IV) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to include Booster Phase.
- ½ (B+OMV) (Group V) Booster Phase: Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation V) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to include Booster Phase.
- PH2 B+OMV (Group VI) Booster Phase: Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation VI) and routine vaccine at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age.
  Group defined to include Booster Phase.
- MenC (Group VII) Booster Phase: Subjects received one dose of meningococcal C conjugate vaccine (Menjugate®; Men C) and routine vaccine at 2,3,4 months of age and one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation VII) and routine vaccine at 12 months of age. One dose of MenC at 13 months of age.
  Group defined to include Booster Phase.
- Par+B+OMV (Group VIII) Booster Phase: Subjects in this group received one dose of meningococcal B recombinant (rMenB) adsorbed vaccine (formulation I) with paracetamol and routine vaccines at 2,3,4,12 months of age and MenC-CRM197 at 13 months of age. Group defined to include Booster Phase.
Arm/Group | B+OMV (Group I) | B+½ OMV (Group II) | B+1/4 OMV (Group III) | B (Group IV) | ½ (B+OMV) (Group V) | PH2 B+OMV (Group VI) | MenC (Group VII) | Par+B+OMV (Group VIII) | B+OMV (Group I) Booster Phase | B+½ OMV (Group II) Booster Phase | B+1/4 OMV (Group III) Booster Phase | B (Group IV) Booster Phase | ½ (B+OMV) (Group V) Booster Phase | PH2 B+OMV (Group VI) Booster Phase | MenC (Group VII) Booster Phase | Par+B+OMV (Group VIII) Booster Phase
Serious Adverse Events (participants affected / at risk) | 16/184 | 20/184 | 12/189 | 20/187 | 13/187 | 16/185 | 11/184 | 15/183 | 14/155 | 7/163 | 12/169 | 5/169 | 15/168 | 9/165 | 9/165 | 14/161
Other Adverse Events (participants affected / at risk) | 181/184 | 183/184 | 186/189 | 183/187 | 180/187 | 180/185 | 175/184 | 175/183 | 151/155 | 159/163 | 162/169 | 152/169 | 154/168 | 156/165 | 155/165 | 150/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B+OMV (Group I) (N=184) | B+½ OMV (Group II) (N=184) | B+1/4 OMV (Group III) (N=189) | B (Group IV) (N=187) | ½ (B+OMV) (Group V) (N=187) | PH2 B+OMV (Group VI) (N=185) | MenC (Group VII) (N=184) | Par+B+OMV (Group VIII) (N=183) | B+OMV (Group I) Booster Phase (N=155) | B+½ OMV (Group II) Booster Phase (N=163) | B+1/4 OMV (Group III) Booster Phase (N=169) | B (Group IV) Booster Phase (N=169) | ½ (B+OMV) (Group V) Booster Phase (N=168) | PH2 B+OMV (Group VI) Booster Phase (N=165) | MenC (Group VII) Booster Phase (N=165) | Par+B+OMV (Group VIII) Booster Phase (N=161)
Cleft palate repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital megacolon (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 3
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myoclonic epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ketosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 4 | 4 | 1 | 2 | 2 | 1 | 1 | 1 | 2 | 0 | 4 | 1 | 3 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 5 | 0 | 3
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bullous impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral myocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acoustic Stimulation Tests (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B+OMV (Group I) (N=184) | B+½ OMV (Group II) (N=184) | B+1/4 OMV (Group III) (N=189) | B (Group IV) (N=187) | ½ (B+OMV) (Group V) (N=187) | PH2 B+OMV (Group VI) (N=185) | MenC (Group VII) (N=184) | Par+B+OMV (Group VIII) (N=183) | B+OMV (Group I) Booster Phase (N=155) | B+½ OMV (Group II) Booster Phase (N=163) | B+1/4 OMV (Group III) Booster Phase (N=169) | B (Group IV) Booster Phase (N=169) | ½ (B+OMV) (Group V) Booster Phase (N=168) | PH2 B+OMV (Group VI) Booster Phase (N=165) | MenC (Group VII) Booster Phase (N=165) | Par+B+OMV (Group VIII) Booster Phase (N=161)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 21 | 9 | 19 | 13 | 19 | 12 | 10 | 5 | 12 | 11 | 9 | 11 | 8 | 10 | 7
Somnolence (Nervous system disorders) | 145 | 149 | 146 | 131 | 142 | 143 | 113 | 134 | 76 | 90 | 90 | 63 | 86 | 88 | 100 | 80
Crying (General disorders) | 122 | 135 | 137 | 99 | 125 | 141 | 87 | 112 | 74 | 64 | 69 | 46 | 71 | 82 | 85 | 50
Injection site erythema (General disorders) | 151 | 150 | 155 | 132 | 131 | 150 | 119 | 132 | 97 | 107 | 120 | 83 | 89 | 96 | 110 | 88
Injection site induration (General disorders) | 141 | 139 | 141 | 126 | 130 | 130 | 122 | 126 | 81 | 90 | 105 | 71 | 76 | 81 | 97 | 70
Injection site pain (General disorders) | 150 | 157 | 139 | 101 | 131 | 152 | 105 | 119 | 121 | 110 | 126 | 92 | 111 | 116 | 125 | 97
Pyrexia (General disorders) | 136 | 127 | 122 | 71 | 114 | 126 | 62 | 78 | 86 | 94 | 70 | 49 | 85 | 72 | 92 | 59
Injection site swelling (General disorders) | 97 | 94 | 103 | 80 | 88 | 100 | 75 | 77 | 57 | 63 | 76 | 46 | 53 | 57 | 65 | 50
Eating disorder (Psychiatric disorders) | 105 | 106 | 104 | 84 | 112 | 119 | 63 | 93 | 74 | 77 | 79 | 52 | 70 | 80 | 72 | 66
Irritability (Psychiatric disorders) | 157 | 159 | 155 | 139 | 151 | 153 | 121 | 137 | 116 | 111 | 112 | 86 | 116 | 115 | 126 | 96
Diarrhoea (Gastrointestinal disorders) | 84 | 87 | 80 | 67 | 80 | 81 | 74 | 73 | 31 | 37 | 39 | 47 | 34 | 31 | 40 | 34
Vomiting (Gastrointestinal disorders) | 38 | 37 | 42 | 32 | 36 | 43 | 34 | 46 | 6 | 13 | 7 | 7 | 10 | 10 | 15 | 20
Dermatitis (Skin and subcutaneous tissue disorders) | 10 | 3 | 7 | 0 | 6 | 2 | 13 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 15 | 18 | 15 | 18 | 24 | 26 | 16 | 19 | 8 | 6 | 11 | 2 | 9 | 6 | 12 | 7
Bronchitis (Infections and infestations) | 34 | 34 | 40 | 31 | 31 | 43 | 34 | 35 | 25 | 18 | 25 | 28 | 28 | 19 | 35 | 17
Conjunctivitis (Infections and infestations) | 14 | 13 | 14 | 13 | 15 | 22 | 10 | 17 | 7 | 7 | 5 | 13 | 8 | 7 | 6 | 10
Ear infection (Infections and infestations) | 10 | 5 | 10 | 6 | 7 | 12 | 9 | 7 | 8 | 4 | 2 | 5 | 9 | 7 | 11 | 4
Exanthema subitum (Infections and infestations) | 9 | 18 | 17 | 17 | 19 | 13 | 20 | 11 | 6 | 7 | 8 | 5 | 5 | 6 | 7 | 10
Gastroenteritis (Infections and infestations) | 10 | 11 | 6 | 9 | 6 | 13 | 7 | 8 | 5 | 4 | 8 | 11 | 12 | 15 | 9 | 7
Nasopharyngitis (Infections and infestations) | 20 | 22 | 25 | 17 | 19 | 24 | 16 | 19 | 15 | 10 | 18 | 11 | 14 | 15 | 14 | 7
Pharyngitis (Infections and infestations) | 21 | 18 | 15 | 21 | 25 | 15 | 18 | 19 | 11 | 16 | 13 | 14 | 22 | 15 | 16 | 15
Rhinitis (Infections and infestations) | 21 | 14 | 12 | 19 | 21 | 26 | 20 | 12 | 7 | 9 | 8 | 11 | 10 | 8 | 6 | 6
Tonsillitis (Infections and infestations) | 6 | 3 | 2 | 12 | 7 | 5 | 5 | 4 | 6 | 10 | 4 | 8 | 5 | 8 | 6 | 9
Upper respiratory tract infection (Infections and infestations) | 13 | 13 | 10 | 10 | 8 | 12 | 9 | 9 | 8 | 7 | 8 | 9 | 7 | 9 | 8 | 5
Varicella (Infections and infestations) | 5 | 10 | 2 | 5 | 7 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 19 | 27 | 23 | 24 | 24 | 17 | 16 | 21 | 12 | 14 | 6 | 16 | 18 | 9 | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days